CLINICAL TRIAL: NCT02848092
Title: Improving ADHD Teen Driving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: St. Louis University (Other); University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01HD084430 (NIH)
Record Dates: First submitted 2016-05-04; First posted 2016-07-28 (Estimated); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Attention Deficit Disorder; Attention Deficit Disorder With Hyperactivity
Keywords: Visual Attention; Automobile Driving
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOCAL+Training (Experimental)
  Interventions: Behavioral: FOCAL+
- Rules of the Road Training (Sham Comparator)
  Interventions: Other: Rules of The road

INTERVENTIONS:
Behavioral: FOCAL+ — Weekly for 5 weeks, teens complete a computer training program designed to train teens to limit the length of glances away from the roadway. On a computer, the top portion of the screen plays a simulated video drive while the bottom half of the screen contains a map. Teens complete tasks that require switching between the 2 halves of the screen. While doing so, they receive feedback regarding how long they are looking away from the driving portion of the screen. After each session of computerized FOCAL training, teens will complete two 5-minute simulated drives. During the drives, teens will be cued to a complete a visual search task which will require them to divert their gaze from the road. Eye tracking goggles will monitor eye glances and provide real time auditory feedback when a visual glance away from the roadway exceeds 2 secs.
  Arms: FOCAL+Training
Other: Rules of The road — Weekly for 5 weeks, teens will perform computer-based training regarding traffic codes, laws, and rules of the road. After each computerized training, teens will complete two 5-minute drives. This time in the driving simulator will be contextualized as a time for them to practice the rules of the road they learned during training. Importantly, teens in the sham intervention group will complete the same distraction tasks but will NOT receive any feedback regarding their eye gaze during simulated driving.
  Arms: Rules of the Road Training

SUMMARY:
Teens with Attention-Deficit/Hyperactivity Disorder (ADHD) have high rates of negative driving outcomes, including motor vehicle crashes, which may be caused by visual inattention (i.e., looking away from the roadway to perform secondary tasks). A driving intervention that trains teens to reduce instances of looking away from the roadway will be tested in teens with ADHD.

DETAILED DESCRIPTION:
Operating a motor vehicle requires a complex set of skills, the most important of which is the ability to continuously visually attend to the roadway. Glances away from the roadway significantly increase one's risk for a motor vehicle crash (MVC). Teen drivers evidence far more extended glances away from the roadway than experienced drivers. Further, teens with a diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD) emit 3-times more extended glances away from the roadway than typical teens. There is a clear need for interventions, particularly one that targets extended glances away from the roadway, to address the driving deficits of teens with ADHD. The proposed research will test the efficacy of the FOcused Concentration and Attention Learning (FOCAL) intervention, which targets reducing the number of extended glances away from the roadway, among teens with ADHD. The PC-based FOCAL training provides teens with an operational understanding of the dangers of extended glances away from the roadway and trains them on limiting the length of the teens' glances. The investigators have enhanced the FOCAL intervention (now termed FOCAL+) to include multiple training sessions and to integrate practice on a driving simulator with immediate feedback regarding extended glance behavior. In this randomized trial, teens with ADHD will be randomly assigned to receive either FOCAL+ or a sham placebo group. Immediately after 1 month of training sessions and 6-months post-training, teens' driving skills will be assessed using a driving simulator. In addition, teens will have cameras installed in their cars for 12-months which record driver behavior and road conditions during irregular events (e.g., hard-braking, swerving). Using data from driving simulation, cameras installed in the teen's car, and teen driving records, the investigators will examine the short- and long-term efficacy of the FOCAL+ intervention on 1) decreasing rates of extended glances away from the roadway among teens with ADHD, and 2) improving driving performance among teens with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16-19.
2. Must meet DSM-5 ADHD criteria for ADHD-Predominantly Inattentive Presentation or ADHD-Combined Presentation based on the K-SADS interview.
3. Possess a valid driver's license and regularly spend at least 3 hours per week engaged in unsupervised driving.
4. IQ ≥80 as measured by the Wechsler Abbreviated Intelligence Scale-II (WASI-II)
5. Parent willing to participate..

Exclusion Criteria:

1. On ADHD medication that cannot be washed out on assessment days.
2. Drug or alcohol dependence according to K-SADS interview.
3. On psychotropic or neuroleptic medications.
4. Require eye glasses (contacts acceptable) for driving (corrective vision restriction on driver's license).

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Epstein, Ph.D, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Center for ADHD, Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Epstein JN, Garner AA, Kiefer AW, Peugh J, Tamm L, MacPherson RP, Simon JO, Fisher DL. Trial of Training to Reduce Driver Inattention in Teens with ADHD. N Engl J Med. 2022 Dec 1;387(22):2056-2066. doi: 10.1056/NEJMoa2204783. PMID 36449421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Teens 16 to 19 years of age with ADHD who had a valid driver's license were recruited at the Cincinnati Children's Hospital Medical Center by means of radio, social media, and print advertisements.
Groups:
- FOCAL+Training: FOCAL+: Weekly for 5 weeks, teens complete a computer training program designed to train teens to limit the length of glances away from the roadway. On a computer, the top portion of the screen plays a simulated video drive while the bottom half of the screen contains a map. Teens complete tasks that require switching between the 2 halves of the screen. While doing so, they receive feedback regarding how long they are looking away from the driving portion of the screen. After each session of computerized FOCAL training, teens will complete up to five 5-minute simulated drives. During the drives, teens will be cued to a complete a visual search task which will require them to divert their gaze from the road. Eye tracking goggles will monitor eye glances and provide real time auditory feedback when a visual glance away from the roadway exceeds 2 secs.
- Rules of the Road Training: Rules of The road: Weekly for 5 weeks, teens will perform computer-based training regarding traffic codes, laws, and rules of the road. After each computerized training, teens will complete up to five 5-minute drives. This time in the driving simulator will be contextualized as a time for them to practice the rules of the road they learned during training. Importantly, teens in the sham intervention group will complete the same distraction tasks but will NOT receive any feedback regarding their eye gaze during simulated driving.
Period: 1-month Post-training Follow-up
Arm/Group | FOCAL+Training | Rules of the Road Training
Started | 76 | 76
Completed | 64 | 71
Not Completed | 12 | 5
Not completed — Lost to Follow-up | 8 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — received new diagnosis of epilepsy | 1 | 0
Not completed — fatigue | 0 | 1
Period: 6-month Post-training Follow-up
Arm/Group | FOCAL+Training | Rules of the Road Training
Started (All randomized participants, irrespective of whether they completed the 1-month post-training follow-up, were recruited to complete the 6-month post-training follow-up.) | 76 | 76
Completed | 63 | 72
Not Completed | 13 | 4
Not completed — Lost to Follow-up | 9 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — frustrated with task | 1 | 0
Not completed — new diagnosis of epilepsy | 1 | 0
Period: 12-month Naturalistic Driving
Arm/Group | FOCAL+Training | Rules of the Road Training
Started (Note that this assessment point reflects 12-months of naturalistic driving beginning at the end of training and ending 1-year post-training.) | 76 | 76
Completed | 73 | 74
Not Completed | 3 | 2
Not completed — Did not have DriveCam installed in car | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOCAL+Training | Rules of the Road Training | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.3 (0.9) | 17.5 (0.9) | 17.4 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 48 | 46 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 75 | 72 | 147
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 65 | 69 | 134
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 76 | 76 | 152
Number of Extended Glances Away from Roadway during Driving Simulation [Mean (Standard Deviation); unit: number of long glances] — Participants completed a simulated drive in a driving simulator with an integrated eye-tracking system. Participants completed two 15-minute drives. During each drive, participants engaged in 14 secondary tasks. The secondary task consisted of searching for streets on a GPS map and lasted for 30 seconds. Eye gaze was sampled continuously. Eye gaze data was summarized by calculating the number of extended (≥2 secs) glances away from the roadway during the 14 secondary task periods per drive. Estimates reflect averages across the 2 drives.
  number of long glances | 21.5 (13.82) | 23.1 (12.28) | 22.43 (13.06)
Standard Deviation of Lateral Position during Driving Simulation [Mean (Standard Deviation); unit: feet] — Participants completed a simulated drive in a driving simulator with an integrated eye-tracking system. Participants completed two 15-minute drives. During each drive, participants engaged in 14 secondary tasks. The secondary task consisted of searching for streets on a GPS map and lasted for 30 seconds. Lateral position was sampled continuously. Standard deviation of lane position was calculated for the 14 secondary task periods per drive. Estimates reflect averages across the 2 drives.
  feet | 1.11 (.33) | 1.20 (.31) | 1.15 (.32)

OUTCOME MEASURES:

1. Primary Outcome: Number of Extended Glances Away From Roadway During Driving Simulation
Description: Participants completed a simulated drive in a driving simulator with an integrated eye-tracking system. Participants completed two 15-minute drives. During each drive, participants engaged in 14 secondary tasks. The secondary task consisted of searching for streets on a GPS map and lasted for 30 seconds. Eye gaze was sampled continuously. Eye gaze data was summarized by calculating the number of extended (≥2 secs) glances away from the roadway during the 14 secondary task periods per drive. This was our primary outcome for visual behavior during driving. Descriptive estimates reflect averages across the 2 drives. However, for analyses, estimates for each drive were statistically modeled with a two-level drive variable.
Time Frame: 1-month post-training
Population: Missing data were handled with the use of 100 imputed data sets that were based on fully conditional specification imputation.
Measure: Mean (95% Confidence Interval); unit: number of long glances
Arm/Group | FOCAL+Training | Rules of the Road Training
Number analyzed (Participants) | 76 | 76
number of long glances | 16.5 [14.0 to 19.1] | 28.0 [26.0 to 30.2]
Statistical Analysis 1: Comparison: FOCAL+Training vs Rules of the Road Training; Test type: Superiority; p < .0001, Generalized Estimating Equation; P value is for the interaction between group (intervention vs. control) and time point (baseline vs. 1 month) using a generalized estimating equation; Incidence Risk Ratio = .64, 95% CI 2-sided [.52 to .76]

2. Primary Outcome: Standard Deviation of Lateral Position During Driving Simulation
Description: Participants completed a simulated drive in a driving simulator with an integrated eye-tracking system. Participants completed two 15-minute drives. During each drive, participants engaged in 14 secondary tasks. The secondary task consisted of searching for streets on a GPS map and lasted for 30 seconds. Lateral position was sampled continuously. Standard deviation of lane position was calculated for the 14 secondary task periods per drive. Estimates reflect averages across the 2 drives. However, for analyses, estimates for each drive were statistically modeled with a two-level drive variable.
Time Frame: 1-month post-training
Population: Missing data were handled with the use of 100 imputed data sets that were based on model-based imputation.
Measure: Mean (95% Confidence Interval); unit: feet
Arm/Group | FOCAL+Training | Rules of the Road Training
Number analyzed (Participants) | 76 | 76
feet | .98 [.92 to 1.04] | 1.20 [1.14 to 1.25]
Statistical Analysis 1: Comparison: FOCAL+Training vs Rules of the Road Training; Test type: Superiority; p < .0001, Generalized Estimating Equation; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -.21, 95% CI 2-sided [-.29 to -.13]

3. Primary Outcome: Number of Extended Glances Away From Roadway During Driving Simulation
Description: as for outcome 1
Time Frame: 6-months post-training
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: number of long glances
Arm/Group | FOCAL+Training | Rules of the Road Training
Number analyzed (Participants) | 76 | 76
number of long glances | 15.7 [13.2 to 18.2] | 27.0 [24.9 to 29.1]
Statistical Analysis 1: Comparison: FOCAL+Training vs Rules of the Road Training; Test type: Superiority; p < .0001, Generalized Estimating Equation; P value is for the interaction between group (intervention vs. control) and time point (baseline vs. 6 month) using a generalized estimating equation; Incidence Risk Ratio = .64, 95% CI 2-sided [.52 to .76]

4. Primary Outcome: Standard Deviation of Lateral Position During Driving Simulation
Description: as for outcome 2
Time Frame: 6-months post-training
Population: Missing data were handled with the use of 100 imputed data sets that were based on model-based imputation.
Measure: Mean (95% Confidence Interval); unit: feet
Arm/Group | FOCAL+Training | Rules of the Road Training
Number analyzed (Participants) | 76 | 76
feet | .98 [.92 to 1.05] | 1.20 [1.14 to 1.27]
Statistical Analysis 1: Comparison: FOCAL+Training vs Rules of the Road Training; Test type: Superiority; p < .0001, Generalized Estimating Equation; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -.22, 95% CI 2-sided [-.31 to -.13]

5. Secondary Outcome: Number of Incidents, Crashes, and Near-crashes Recorded With DriveCam
Description: The DriveCam device is an event-triggered palm sized pair of cameras that are mounted to the rear view mirror of the participant's car. The device has a forward-road facing camera and another camera that faces the driver. Both cameras continuously record but only save to memory when a built-in accelerometer exceeds a set g force threshold. Any g-force event that exceeds .6 g-force will be coded using codings of crashes (i.e., collision with another vehicle or object) or near-crashes (i.e., an evasive maneuver performed to avoid a MVC). This outcome will include the rate of crashes or near-crashes.
Time Frame: 12 months
Population: These analyses were conducted in the as-treated population, which involved participants for whom data from the in-vehicle recording device were available. Three teens (1 in the intervention group and 2 in the control group) had no g-force events during the 1-year follow-up for the evaluation of secondary outcomes.
Measure: Count of Units; unit: DriveCam events
Units Other Than Participants: DriveCam events
Arm/Group | FOCAL+Training | Rules of the Road Training
Number analyzed (Participants) | 72 | 72
Number analyzed (DriveCam events) | 3213 | 2818
DriveCam events | 110 | 159
Statistical Analysis 1: Comparison: Rules of the Road Training; Test type: Superiority; Risk Ratio (RR) = .60, 95% CI 2-sided [.41 to .89]

6. Secondary Outcome: Number of DriveCam Events That Are Preceded by a 2 Second or Greater Glance Away From the Roadway
Description: The DriveCam device has a forward-road facing camera and another camera that faces the driver. Both cameras record when a built-in accelerometer exceeds a set g force threshold of .6. Video event recordings of the driver were be coded for whether a 2-second or longer glance away from the roadway occurred during the recorded event. Using these codings, the number of events that included a 2-second or longer glance away from the roadway was determined for each group.
Time Frame: 12 months
Population: as for outcome 5
Measure: Count of Units; unit: DriveCam events
Units Other Than Participants: DriveCam events
Arm/Group | FOCAL+Training | Rules of the Road Training
Number analyzed (Participants) | 72 | 72
Number analyzed (DriveCam events) | 3213 | 2818
DriveCam events | 588 | 674
Statistical Analysis 1: Comparison: Rules of the Road Training; Test type: Superiority; Risk Ratio (RR) = .76, 95% CI 2-sided [.61 to .92]

ADVERSE EVENTS:
Time Frame: 5-weeks of training, 1-month post-training assessment, 6-month post-training assessment
Description: Anticipated AE and possible precautions and responses to these events include: 1) Simulator sickness including nausea and headache. 2) Frustration with simulator training.
Arm/Group | FOCAL+Training | Rules of the Road Training
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 8/76 | 6/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOCAL+Training (N=76) | Rules of the Road Training (N=76)
Simulator sickness during assessment (Nervous system disorders) | 0 (0) | 2 (2)
Simulator sickness during training (Nervous system disorders) | 6 (6) | 4 (4)
Frustration during training (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT02848092/Prot_SAP_000.pdf
  • Informed Consent Form: Parent Permission Form (2019-03-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT02848092/ICF_001.pdf
  • Informed Consent Form: Adult Consent Form (2019-03-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT02848092/ICF_002.pdf